CLINICAL TRIAL: NCT05460806
Title: The Effect of Aerobic Exercise on Pain, Alexithymia Level and Quality of Life in Alexithymic Individuals With Chronic Pain
Brief Title: The Effect of Aerobic Exercise in Alexithymic Individuals With Chronic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KTO Karatay University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KaratayUH5
Record Dates: First submitted 2022-07-13; First posted 2022-07-15 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-07

CONDITIONS: Chronic Pain; Quality of Life; Alexithymia
MeSH Terms: conditions — Chronic Pain; Affective Symptoms | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic Exercise (Experimental): Participants assigned to aerobic exercise training will walk on a treadmill (RodbyTM, RL 1600E, Enhorna, Sweden) for 40 minutes at an intensity of 60-75% of maximum heart rate (220-age formula) three times per week for 8 weeks. The heart rate of the participants will be measured with an electric heart rate monitor throughout the session.
  Interventions: Other: Aerobic Exercise
- Control (No Intervention)

INTERVENTIONS:
Other: Aerobic Exercise — Participants assigned to aerobic exercise training will walk on a treadmill (RodbyTM, RL 1600E, Enhorna, Sweden) for 40 minutes at an intensity of 60-75% of maximum heart rate (220-age formula) three times per week for 8 weeks. The heart rate of the participants will be measured with an electric heart rate monitor throughout the session.
  Arms: Aerobic Exercise

SUMMARY:
It was aimed to investigate the effect of aerobic exercise on pain, alexithymia level and quality of life in young alexithymic individuals with chronic pain. There is no study in the literature comparing the effectiveness of aerobic exercise on alexithymia and chronic pain. Since our study will be the first study to investigate the subject, we foresee that it is scientifically important and will shed light on future studies. In addition, it is planned to make national or international papers and publications after the study is completed.

DETAILED DESCRIPTION:
In the study, after the necessary permissions are obtained, the Graded Chronic Pain Scale (ECAS) and Toronto Alexithymia Scale-20 (TAS-20) will be sent to the students who are studying at KTO Karatay University and whose age range is between 18-25 years. Among the students who fill out the form voluntarily, individuals who mark the 3rd or 4th option in the first question in the DKAS and who have a total score of 52 and above in the TAS-20 scale will be identified. Among these individuals, a total of 40 people will be included in the study randomly with a computer program. These participants will again be randomly divided into two groups as the control group (n=20) and the exercise group (n=20).

ELIGIBILITY:
Inclusion Criteria:

* To be between the ages of 18-25
* To mark the 3rd or 4th option in the first question in the DKAS
* To have a TAS-20 total score of 61 and above

Exclusion Criteria:

* Presence of any physiological or psychological disease that may interfere with the exercise protocol to be applied

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2022-07-12 (Actual); Primary Completion 2022-09-06 (Actual); Study Completion 2022-09-07 (Actual)

PRIMARY OUTCOMES:
Alexithymia | Change from Baseline Alexithymia after 8 week exercise
  Alexithymia levels will be assessed on the Toronto Alexithymia Scale-20 before and after work.

SECONDARY OUTCOMES:
Pain levels | Change from Baseline pain after 8 week exercise
  Pain levels will be assessed on the VAS before and after work.
Quality of Life levels | Change from Baseline quality of life after 8 week exercise
  Quality of life levels will be assessed on the SF36 before and after work.

CONTACTS AND LOCATIONS:
Locations (1):
- KTO Karatay University, Konya, Karatay, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No